CLINICAL TRIAL: NCT07281820
Title: FRAME (Focused Recognition, Assessment and Management of Late Effects): A Single-Center Implementation Study Using RE-AIM to Guide Evaluation in the Department of Oncology, Vejle Hospital
Brief Title: FRAME - Implementation of a PRO Measure to Inform Patient-Centered Survivorship Care in Oncology Outpatient Visits
Acronym: FRAME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: FRAME-PRO; R392-A23403 (Other Grant/Funding Number: Danish Cancer Society)
Record Dates: First submitted 2025-11-14; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Cancer; Late Effects
Keywords: Patient-reported outcomes; Survivorship; Oncology; Implementation science; RE-AIM; Proctor Outcomes; Stepped-care
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm - Department-wide implementation of FRAME (Other): FRAME model (questionnaire + dialogue + management plan)
  Interventions: Behavioral: FRAME model (questionnaire + dialogue + management plan)

INTERVENTIONS:
Behavioral: FRAME model (questionnaire + dialogue + management plan) — Administration of the patient-developed FRAME-PRO prior to the visit; clinician-patient dialogue guided by responses; stepped-care management/referrals; documentation via standard EHR phrase. Implementation strategies include educational meetings/materials, ongoing training, audit & feedback at weekly huddles, reminders/prompts, local champions, and local technical assistance.

SUMMARY:
FRAME is a patient-centered survivorship care model embedded in routine oncology visits. It consists of: (1) a pre-visit patient-reported questionnaire (FRAME-PRO), (2) a clinician-patient dialogue guided by the responses, and (3) a tailored management plan including stepped-care referrals (general practitioner and municipality; oncology department supportive services; specialized late-effects clinics). The implementation is evaluated with the RE-AIM framework supplemented by Proctor implementation outcomes. Data sources include the "Mit Sygehus" app, departmental registries, purpose-built questionnaires, fidelity checklists, and qualitative interviews with clinicians, patients, and informal caregivers.

DETAILED DESCRIPTION:
The project implements FRAME at the Department of Oncology, Vejle Hospital. The FRAME-PRO enables patients and informal caregivers to reflect on late effects and needs before the visit. During the visit, clinicians access FRAME-PRO electronically to prioritize what matters most, assess severity (triage), and co-create a management plan documented in the electronic health record using a purpose-developed standard phrase to support cross-sector information transfer. Implementation strategies are informed by the Expert Recommendations for Implementing Change (ERIC) and local logs (education, audit & feedback, reminders, local champions, technical assistance). Evaluation follows RE-AIM: Reach (completion of FRAME-PRO), Effectiveness (referrals to supportive care, quality of life, time use), Adoption (clinician use), Implementation (fidelity to opening, discussing, and managing needs), and Maintenance (sustained use). Quantitative data are summarized descriptively; qualitative data are analyzed with content analysis. Ethics approval covers interviews with patients, caregivers, and clinicians.

ELIGIBILITY:
Inclusion Criteria:

- All oncologists conducting outpatient visits at the Department of Oncology, Vejle Hospital during the study period.

Exclusion Criteria:

- None.

Participants for interviews:

* A purposive sample of patients, informal caregivers, and clinicians approached ≥6 months after launch
* written and verbally informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of oncologists who actively use FRAME in ≥50% of eligible outpatient visits. | 3 months
  Adoption

SECONDARY OUTCOMES:
Proportion of eligible outpatient visits with completed FRAME-PRO (via "Mit Sygehus"). | Continuously during implementation (up to 6 months)
  Reach
Change in proportion of visits/patients with referrals to supportive care units compared with pre-implementation baseline. | Up to 6 months
  Effectiveness. Target: +15% (exploratory).
Change in patient-reported global quality of life measured on a Likert-like scale from 1 (poor) to 5 (excellent). | Up to 6 months
  Effectiveness. Target: +10% relative increase (exploratory).
Degree to which clinicians and patients (a) open FRAME-PRO during the visit (yes/no), (b) discuss reported needs (yes/no), and (c) manage needs aligned with preferences (yes/no) | Up to 6 months
  Implementation / fidelity
Perceived feasibility of active FRAME use among clinicians on a likert-like scale from 1 (not feasible) to 5 (very feasible) | 6 months
  Feasibility of FRAME (Proctor outcome)
Clinician-perceived acceptability of FRAME-supported visits on a scale from 1 (not acceptable) to 5 (very acceptable) | 6 months
  Acceptability (Proctor outcome)
Perceived fit of FRAME to the oncology outpatient setting and patient population on a scale from 1 (not appropriate) to 5 (very appropriate). | 6 months
  Appropriateness (Proctor outcome)
Time needed to include FRAME-PRO in the visit on a scale from 1 (definitely shorter time with FRAME) to 5 (definitely longer time with FRAME). | 6 months
  Cost
Integration of FRAME within the outpatient clinic (e.g., percent of clinicians using FRAME routinely) | 6 months
  Penetration
Sustained active use of FRAME among clinicians in the last 3 months of the study window. | Up to 12 months
  Maintenance
Proportion of patients referred to supportive care units (actual numbers) | 6 months
  Effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: Torben F Hansen, Dr. Med., Study Director — Department of Oncology, Vejle Hospital, University Hospital of Southern Denmark, Denmark
Locations (1):
- Department of Oncology, Vejle Hospital, University Hospital of Southern Denmark, Vejle, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lyhne JD, Gade L, Hansen L, Johansen A, Smith A', Jensen LH, Ventzel L. Survivor-driven development of a PROM for use in routine colorectal cancer care. Acta Oncol. 2025 Mar 27;64:475-483. doi: 10.2340/1651-226X.2025.42032. PMID 40150842